CLINICAL TRIAL: NCT06739044
Title: A Multicenter, Randomized, Open-label, Parallel-controlled Phase III Clinical Study Comparing the Efficacy and Safety of Semaglutide Injection With Ozempic ® in Patients With Type 2 Diabetes Mellitus Who Have Inadequate Glycemic Control With Metformin
Brief Title: Efficacy and Safety of Semaglutide Injection vs Ozempic® in Patients With Type 2 Diabetes
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Hangzhou Zhongmei Huadong Pharmaceutical Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: HDG1901-301
Record Dates: First submitted 2024-12-10; First posted 2024-12-18 (Actual); Last update posted 2025-07-28 (Actual); Status verified 2024-12

CONDITIONS: Type 2 Diabetes
Keywords: Glucagon-Like Peptide-1 Receptor Agonists; semaglutide
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — semaglutide

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Experimental group (Experimental)
  Interventions: Drug: HDG1901
- Active Comparator (Active Comparator)
  Interventions: Drug: Ozempic®

INTERVENTIONS:
Drug: Ozempic® — The starting dose is 0.25 mg once weekly. After 4 weeks the dose should be increased to 0.5 mg once weekly. After at least 4 weeks with a dose of 0.5 mg once weekly, the dose can be increased to 1 mg once weekly for 24 weeks.
  Arms: Active Comparator
Drug: HDG1901 — The starting dose is 0.25 mg once weekly. After 4 weeks the dose should be increased to 0.5 mg once weekly. After at least 4 weeks with a dose of 0.5 mg once weekly, the dose can be increased to 1 mg once weekly for 24 weeks.
  Arms: Experimental group

SUMMARY:
This is a 32-week randomized, open-label, parallel-controlled biosimilar comparison study comparing the efficacy, safety and immunogenicity of the investigational drug and the active comparator in patients with type 2 diabetes mellitus who have inadequate glycemic control with metformin. Eligible participants will be screened and randomized to the experimental group and the active comparator group at a ratio of 1:1 , semaglutide injection or Ozempic® injection abdominal subcutaneous injection will be given according to their groups weekly for 32 weeks. Follow-up for 4 weeks after administration.

Trial product will be add-on to subject's stable pre-trial metformin.

The study included a screening period (up to 2 weeks), run-in period（6 weeks），baseline, administration period(32 weeks), and a follow-up period (4 weeks). The duration of the study will be approximately 44 weeks for a participant.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female, age 18-75 years (both inclusive) at the time of signing informed consent
2. Subjects diagnosed with type 2 diabetes and on stable treatment in a period of 6 weeks prior to screening with metformin ≥ 1500 mg (or maximum tolerated dose ≥ 1000 mg)
3. HbA1c 7.5 - 11.0 % (both inclusive) (screening)
4. HbA1c 7.0 - 10.5 % (both inclusive) (randomisation)
5. BMI 18.5-35 kg/m2 (both inclusive)

Exclusion Criteria:

1. Other types of diabetes besides Type 2 diabetes
2. A history of acute diabetes complications within 6 months before screening
3. A history of acute or chronic pancreatitis, symptomatic gallbladder disease, or other high-risk factors that may lead to pancreatitis
4. Personal or family history of medullary thyroid cancer (MTC) or multiple endocrine neoplasia syndrome type 2 (MEN 2)
5. Acute coronary or cerebrovascular event within 3 months before screening or randomisation
6. Heart failure, New York Heart Association (NYHA) class IV
7. Treatment with glucose lowering agent(s) other than stated in the inclusion criteria in a period of 6 weeks before screening. An exception is short-term treatment (≤7 days in total) with insulin in connection with inter-current illness
8. Fasting Plasma Glucose (FPG) ≥ 13.9mmol/L
9. Screening calcitonin value ≥ 35 ng/L (pg/mL)
10. Estimated glomerular filtration rate (eGFR) < 60 ml/min/1.73 m2
11. Any disorder which, in the opinion of the investigator, might jeopardise subject's safety or compliance with the protocol

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 494 (Actual)
Dates: Start 2023-09-20 (Actual); Primary Completion 2024-10-11 (Actual); Study Completion 2025-02-21 (Actual)

PRIMARY OUTCOMES:
Change in HbA1c from baseline | Week 32

SECONDARY OUTCOMES:
Change in HbA1c from baseline | Week 20
Change in Fasting Plasma Glucose(FPG) from baseline | Week 20， Week 32
HbA1c ≤ 6.5% | Week 20, Week 32
HbA1c ≤ 7.0% | Week 20，Week 32
C-peptide | Week 20, Week 32
Insulin | Week 20, Week 32

CONTACTS AND LOCATIONS:
Locations (1):
- Beijing Hospital, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: No